CLINICAL TRIAL: NCT04855617
Title: Symptom Burden in Patients Treated With Ocrelizumab for Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-00041
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Study-specific biospecimens (peripheral venous blood) will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients Receiving Multiple Sclerosis care: Patients currently receiving ocrelizumab or initiating ocrelizumab per their MS treating physician.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Administer Ocrelizumab under the close supervision of an experienced healthcare professional with access to appropriate medical support to manage severe reactions such as serious infusion reactions.
  * Initial dose: 300 mg intravenous infusion, followed two weeks later by a second 300 mg intravenous infusion.
  * Subsequent doses: single 600 mg intravenous infusion every 6 months.
  * Observe the patient for at least one hour after the completion of the infusion
  Other Names: OCREVUS

SUMMARY:
This study is designed to determine whether symptom burden differs by time to infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Diagnosis of multiple sclerosis (revised 2017 criteria)
* EDSS 0-7
* Plans to initiate treatment with ocrelizumab within 6 months or has been on an approved regimen of ocrelizumab for >12 months as part of their clinical care
* Individual must be able to provide consent, read/write/comprehend English Language

Exclusion Criteria:

* Clinical relapse within 3 months of first on-study infusion
* Cognitive impairment limiting the ability to consent or fill out the electronic survey
* Currently pregnant, planning to become pregnant during the study period, or currently breastfeeding
* Untreated psychiatric illness (such as major depressive disorder, Bipolar disorder, psychotic disorder, schizophrenia)
* Active substance abuse disorder
* Significant medical comorbidities (such as history of severe traumatic brain injury, stroke, systemic cancer or chronic infection)
* Chemotherapy use within 6 months of first study infusion
* Prior treatment with alemtuzumab within 12 months of first study infusion
* Prior treatment with a B-cell depleting therapy other than ocrelizumab within 12 months of first on-study infusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving Multiple Sclerosis care at the NYU Comprehensive MS Care Center or the Elliot Lewis MS Center will be recruited. A clinical list of patients currently receiving ocrelizumab, or potentially starting ocrelizumab will be screened for study inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life in Neurologic Disorders (NeuroQoL) Scores | Week 4, Week 22
  The NeuroQoL short form will be used for this study, which consists of 5 statements on how much difficulty one currently has during certain activities. Each statement is answered on a scale of 1 (cannot do) to 5 (none); the total range of score is 1-25. The higher the score, the less difficulty one has.

SECONDARY OUTCOMES:
Change in SymptoMScreen (SyMS) Scores | Week 4, Week 22
  SyMS consists of 12 questions. Participants are asked to choose a response that best describes how each MS symptom has affected everyday life activities. Each questions is answered on a scale of 0 (not affected at all) to 6 (total limitation/I'm unable to do most daily activities); the total range of score is 0-72. The higher the score, the higher the limitation from MS symptoms.
Change in Work Productivity and Activity Impairment Questionnaire: MS (WPAI:MS) Scores | Week 4, Week 22
  There are 2 questions that are quantifiable - they pertain to how much MS has affected one's productivity while working or ability to do regular daily activities. The questions are answered on a scale of 0 (no effect) to 10 (complete prevention); the total range of score is 0-20. The higher the score, the higher the level of prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Kister, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Elliot Lewis Center for Multiple Sclerosis Care, Wellesley, Massachusetts
  - NYU Langone Health Multiple Sclerosis Comprehensive Care Center (NYULH MSCCC), New York, New York